CLINICAL TRIAL: NCT06264648
Title: Investigation of Palpation Pressure Sensitivity of Physiotherapists
Brief Title: Investigation of Palpation Pressure Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ömer Osman Pala, Associated Professor Doctor, Abant Izzet Baysal University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AIBU-FTR-OOP-04
Record Dates: First submitted 2023-11-14; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Sensitivity Training Groups
Keywords: Palpation; Manual therapy; Pressure

STUDY DESIGN:
Intervention Model Description: 2 groups of physiotherapists with different fields of experience were attended to study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy using group (Experimental): This group includes physiotherapists that using manual therapy techniques.
  Interventions: Other: Pressure sensitivity education
- Non Manual Therapy using (Experimental): This group includes physiotherapists using different techniques during working, not manual therapy
  Interventions: Other: Pressure sensitivity education

INTERVENTIONS:
Other: Pressure sensitivity education — Therapists were asked to apply pressure to the scale with estimated weights of 0.5 kg, 1 kg, 2 kg and 4 kg. In each measurement, the value shown on the scale was recorded without being shown to the participant.After the measurements, the participants were made to experiment when the digital screen can be seen, in order to teach the physiotherapists how much pressure they applied to reach the target weight. Participants were given a total of 10 minutes for the trials. Then, the digital screen was hidden again, and the therapist was asked to apply 0.5 kg, 1 kg, 2 kg and 4 kg weight in a randomized order and maintain this pressure for 5 seconds. The weight fixed by the therapist for 5 seconds was noted by the researcher; the participant was not informed about the values on the digital screen.

SUMMARY:
The study is planned for searching physiotherapists palpation abilities. There were 2 groups of physiotherapists. They were asked for to push target pressures. After making some exercise, the assesment was done again.

DETAILED DESCRIPTION:
2 groups of physiotherapists with different fields of experience were attended to study. Fingers are positioned on the marked area at the center point of the scale. Therapists were asked to apply pressure to the scale with estimated weights of 0.5 kg, 1 kg, 2 kg and 4 kg. In each measurements, the value on the scale was recorded without being shown to the participants. After the measurements, the participants were made to experiment when the digital screen can be seen, in order to teach the physiotherapists how much pressure they applied to reach the target weight. Participants were given a total of 10 minutes for the trials. Then, the digital screen was hidden again, and the therapist was asked to apply 0.5 kg, 1 kg, 2 kg and 4 kg weight in a randomized order and maintain that pressure for 5 seconds. The weight fixed by the therapist for 5 seconds was noted by the researcher; the participant was not informed about the values on the digital screen.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate,
* Active working patients as a physiotherapists pediatric, neurologic, orthopedic physiotherapy, manual therapy or osteopathy.

Exclusion Criteria:

* Having a neurological disease (multiple sclerosis, polyneuropathy, etc.) -Having a disease that may cause neurological deficit in the upper extremity (cervical myelopathy, carpal tunnel syndrome, pronator teres syndrome, cubital tunnel syndrome, ---
* Guyon canal syndrome)
* Refuse to participate

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Measurement Palpation Pressure with Digital Scale | baseline
  The digital scale will used to assess the palpation pressure of participants. This digital scale is designed for a measurement range of 1-10.000 gr. Palpation pressures will measure at baseline and after education to see whether any changes.
Measurement Palpation Pressure with Digital Scale | 10 minute after pressure sensitivity education
  The digital scale will used to assess the palpation pressure of participants. This digital scale is designed for a measurement range of 1-10.000 gr. Palpation pressures will measure at baseline and after education to see whether any changes.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Osman Pala, Assoc. Prof, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Faculty of Health Sciences Bolu Abant İzzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No